CLINICAL TRIAL: NCT07319104
Title: Biobank for Validating Liquid Biopsy in Predicting the Prognosis of Superficial Colonic Lesions
Brief Title: Liquid Biopsy in Early Colorectal Lesions
Acronym: FECCO-BioBank
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Limoges (Other); Société Nationale Française de Gastroentérologie (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL25_0092; 2025-A02328-41 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2025-12-02; First posted 2026-01-06 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Neoplasms; Precancerous Conditions; Adenocarcinoma of the Colon; Lymphatic Metastasis; Endoscopy, Gastrointestinal; Liquid Biopsy; Biomarkers
MeSH Terms: conditions — Colorectal Neoplasms; Precancerous Conditions; Colonic Neoplasms; Lymphatic Metastasis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Blood samples will be taken before and after submucosal dissections, processed, and then stored as plasma. Further in-depth analyses can then be performed, including analyses of circulating tumor DNA, broad protein panels, exosomes, extracellular vesicles, and immune system cells, etc.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Venous blood sampling — Five 6-7 ml EDTA tubes of venous blood will be collected at two points during the care pathway:
  * Immediately before the endoscopic procedure, at the time of catheter insertion for general anesthesia. This is to study the signal intensity at a baseline stage.
  * Between 2 and 6 weeks after submucosal dissection (only in cases of pT1 adenocarcinoma) and before any further surgery for pT1 cancer. This is to study the presence or absence of a residual signal after local resection.
  Other Names: Blood sample

SUMMARY:
Early colorectal cancer screening increasingly detects small superficial colonic lesions, but current diagnostic tools still struggle to distinguish benign from malignant lesions and to assess lymph node risk. As histology after resection has limited accuracy, many patients undergo unnecessary surgery.

Liquid biopsy, analyzing circulating biomarkers such as tumor DNA, extracellular vesicles, and nucleosomes, offers a non-invasive way to better classify these lesions. Emerging evidence suggests it may outperform current criteria for predicting lymph node involvement in T1 colorectal cancer.

This study will establish a biobank of 1,000 patients to identify blood-based signatures that predict tumor stage and lymph node status. The hypothesis of the study is that circulating biomarkers can accurately differentiate benign from malignant lesions and identify patients with or without lymph node metastasis.

DETAILED DESCRIPTION:
Introduction :

Early colorectal cancer screening increasingly identifies superficial colonic lesions, but current diagnostic tools often fail to accurately distinguish benign from malignant lesions or to predict lymph node involvement. As histological criteria have limited predictive value, many patients with T1 tumors undergo unnecessary surgery. Liquid biopsy, based on circulating blood biomarkers, offers a promising non-invasive alternative that may improve diagnostic precision.

Aim :

The study aims to build a biobank of 1,000 patients with superficial colonic tumors to identify and validate circulating biomarker signatures capable of predicting tumor malignancy and lymph node status. The hypothesis is that liquid biopsy markers can reliably differentiate benign from malignant lesions and identify patients at risk of lymph node metastasis.

Methods :

This is a multicenter prospective cohort study embedded in the FECCo cohort. Blood samples will be collected at the time of endoscopic resection and, for pT1 lesions, again 2-6 weeks later. Clinical data will be retrieved annually from the FECCo database. Diagnostic performance of circulating biomarkers will be assessed using ROC curves, logistic regression (Lasso), and bootstrap validation to identify signatures associated with malignancy and lymph node involvement.

ELIGIBILITY:
Inclusion Criteria:

* Patient of legal age (≥ 18 years)
* Patient with a superficial colonic tumor treated by submucosal dissection
* Patient included in the FECCo cohort
* Patient wishing to participate in the FECCO-BioBank biological collection

Exclusion Criteria:

* Person with significant comorbidities preventing blood sampling
* Patients with a distant metastasis detected by imaging
* Person unable to read and write French
* Person who have expressed their opposition to participating in this research after being informed by an investigator and having read the information sheet
* Person not benefiting from a national health insurance scheme
* Person under legal protection, guardianship or curatorship
* Person participating in other study with an ongoing exclusion period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be identified and recruited in gastroenterology consultations, within the investigating centers to which they will be referred as part of routine care.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Extracellular vesicles (EVs) | Morning of endoscopic resection (Day 0), 2 and 6 weeks after Day 0 (only for pT1 tumor)
  Detection of plasma extracellular vesicles (EVs):
  * to predict the presence of adenocarcinomatous degeneration (malignant profile) vs. dysplasia (benign profile)
  * to differentiate patients with pT1 adenocarcinoma of the colon, with lymph node metastasis (N+), from those without lymph node metastasis (N-) before treatment.

SECONDARY OUTCOMES:
Circulating nucleosomes | Morning of endoscopic resection (Day 0), 2 and 6 weeks after Day 0 (only for pT1 tumor)
  Detection of circulating nucleosomes:
  * to predict the presence of adenocarcinomatous degeneration (malignant profile) vs. dysplasia (benign profile)
  * to differentiate patients with pT1 adenocarcinoma of the colon, with lymph node metastasis (N+), from those without lymph node metastasis (N-) before treatment.
Circulating tumor DNA (ctDNA) | Morning of endoscopic resection (Day 0), 2 and 6 weeks after Day 0 (only for pT1 tumor)
  Detection of ctDNA:
  * to predict the presence of adenocarcinomatous degeneration (malignant profile) vs. dysplasia (benign profile)
  * to differentiate patients with pT1 adenocarcinoma of the colon, with lymph node metastasis (N+), from those without lymph node metastasis (N-) before treatment.
Circulating proteomic profile via O-link technology | Morning of endoscopic resection (Day 0), 2 and 6 weeks after Day 0 (only for pT1 tumor)
  Detection of circulating proteomic profile via O-link technology:
  * to predict the presence of adenocarcinomatous degeneration (malignant profile) vs. dysplasia (benign profile)
  * to differentiate patients with pT1 adenocarcinoma of the colon, with lymph node metastasis (N+), from those without lymph node metastasis (N-) before treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine DEBOURDEAU, MD, Study Chair — University Hospital, Montpellier
Locations (12):
- France (12):
  - University Hospital of Amiens, Amiens
  - University Hospital of Bordeaux, Bordeaux
  - University Hospital of Brest, Brest
  - University Hospital of Dijon, Dijon
  - University Hospital of Limoges, Limoges
  - Civil Hospices of Lyon, Lyon
  - Jean Mermoy Private Hospital, Lyon
  - University Hospital of Montpellier, Montpellier
  - University Hospital of Nancy, Nancy
  - University Hospital of Nîmes, Nîmes
  - Saint Joseph Hospital, Paris
  - University Hospital of Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lecomte T, Tougeron D, Chautard R, Bressand D, Bibeau F, Blanc B, Cohen R, Jacques J, Lagasse JP, Laurent-Puig P, Lepage C, Lucidarme O, Martin-Babau J, Panis Y, Portales F, Taieb J, Aparicio T, Bouche O; Thesaurus National de Cancerologie Digestive (TNCD); Societe Nationale Francaise de Gastroenterologie (SNFGE); Federation Francophone de Cancerologie Digestive (FFCD); Groupe Cooperateur multidisciplinaire en Oncologie (GERCOR); Federation Nationale des Centres de Lutte Contre le Cancer (UNICANCER); Societe Francaise de Chirurgie Digestive (SFCD); Societe Francaise d'Endoscopie Digestive (SFED); Societe Francaise de Radiotherapie Oncologique (SFRO); Association de Chirurgie Hepato-Bilio-Pancreatique et Transplantation (ACHBT); Societe Francaise de Pathologie (SFP); Association Francaise pour l'Etude du Foie (AFEF); Societe Francaise de Radiologie (SFR). Non-metastatic colon cancer: French Intergroup Clinical Practice Guidelines for diagnosis, treatments, and follow-up (TNCD, SNFGE, FFCD, GERCOR, UNICANCER, SFCD, SFED, SFRO, ACHBT, SFP, AFEF, and SFR). Dig Liver Dis. 2024 May;56(5):756-769. doi: 10.1016/j.dld.2024.01.208. Epub 2024 Feb 20. PMID 38383162
- [Background] Zwager LW, Bastiaansen BAJ, Montazeri NSM, Hompes R, Barresi V, Ichimasa K, Kawachi H, Machado I, Masaki T, Sheng W, Tanaka S, Togashi K, Yasue C, Fockens P, Moons LMG, Dekker E. Deep Submucosal Invasion Is Not an Independent Risk Factor for Lymph Node Metastasis in T1 Colorectal Cancer: A Meta-Analysis. Gastroenterology. 2022 Jul;163(1):174-189. doi: 10.1053/j.gastro.2022.04.010. Epub 2022 Apr 15. PMID 35436498
- [Background] Alix-Panabieres C, Pantel K. Liquid Biopsy: From Discovery to Clinical Application. Cancer Discov. 2021 Apr;11(4):858-873. doi: 10.1158/2159-8290.CD-20-1311. PMID 33811121
- [Background] Chung DC, Gray DM 2nd, Singh H, Issaka RB, Raymond VM, Eagle C, Hu S, Chudova DI, Talasaz A, Greenson JK, Sinicrope FA, Gupta S, Grady WM. A Cell-free DNA Blood-Based Test for Colorectal Cancer Screening. N Engl J Med. 2024 Mar 14;390(11):973-983. doi: 10.1056/NEJMoa2304714. PMID 38477985
- [Background] Wada Y, Shimada M, Murano T, Takamaru H, Morine Y, Ikemoto T, Saito Y, Balaguer F, Bujanda L, Pellise M, Kato K, Saito Y, Ikematsu H, Goel A. A Liquid Biopsy Assay for Noninvasive Identification of Lymph Node Metastases in T1 Colorectal Cancer. Gastroenterology. 2021 Jul;161(1):151-162.e1. doi: 10.1053/j.gastro.2021.03.062. Epub 2021 Apr 2. PMID 33819484
- [Background] Miyazaki K, Wada Y, Okuno K, Murano T, Morine Y, Ikemoto T, Saito Y, Ikematsu H, Kinugasa Y, Shimada M, Goel A. An exosome-based liquid biopsy signature for pre-operative identification of lymph node metastasis in patients with pathological high-risk T1 colorectal cancer. Mol Cancer. 2023 Jan 6;22(1):2. doi: 10.1186/s12943-022-01685-8. PMID 36609320
- [Background] Schlemper RJ, Riddell RH, Kato Y, Borchard F, Cooper HS, Dawsey SM, Dixon MF, Fenoglio-Preiser CM, Flejou JF, Geboes K, Hattori T, Hirota T, Itabashi M, Iwafuchi M, Iwashita A, Kim YI, Kirchner T, Klimpfinger M, Koike M, Lauwers GY, Lewin KJ, Oberhuber G, Offner F, Price AB, Rubio CA, Shimizu M, Shimoda T, Sipponen P, Solcia E, Stolte M, Watanabe H, Yamabe H. The Vienna classification of gastrointestinal epithelial neoplasia. Gut. 2000 Aug;47(2):251-5. doi: 10.1136/gut.47.2.251. PMID 10896917